CLINICAL TRIAL: NCT04824612
Title: Effect of the Combination of Photobiomodulation Therapy and the Intralesional Administration of Corticoid in the Preoperative and Postoperative Periods of Keloid Surgery: a Randomized, Controlled, Double-blind Trial
Brief Title: Photobiomodulation and the Intralesional Administration of Corticoid in the Keloid Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, CLINICAL PROFESSOR, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Keloid
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Keloid; Cicatrix
Keywords: keloid; photobiomodulation; corticoid
MeSH Terms: conditions — Keloid; Cicatrix | interventions — Low-Level Light Therapy; triamcinolone hexacetonide

STUDY DESIGN:
Intervention Model Description: 58 patients will be allocated in the experimental and control groups: sham (N = 29): intralesional administration of corticoid (IAC) and sham PBM in the preoperative and postoperative periods of keloid removal surgery; and experimental group with active PBM combined with IAC (N = 29) in the preoperative and postoperative periods of keloid removal surgery. Transcutaneous PBM will be performed on the keloid in the preoperative period and on the remaining scar in the postoperative period using blue LED (470 nm, 0,4 W, 24J per point on 10 linear points, total 240J).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The evaluator, analyst, and participants will be unaware of the group to which the participants are allocated. The operator will also be unaware of whether the blue light has a biological effect or is a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Group (Sham Comparator): intralesional administration of corticoid (IAC): intralesional injection of 20 mg/ml triamcinolone hexacetonide (Triancil®, Apsen Farmacêutica S.A.) - two injections in the preoperative period with a two-week interval between injections and a monthly injection for three months in the postoperative period. The injections will be intralesional and will not surpass the dermis. The drug will be diluted with the same quantity of 2% lidocaine. The scar will be divided into equal parts of 1 cm² and the drug will be distributed equally, respecting the total dose per session of 20 mg for the face and 40 mg for other topographies.
  Sham PBM in the preoperative and postoperative periods of keloid removal surgery: Preoperative: every two weeks for 30 days. Postoperative: Immediately after surgery, weekly for 4 weeks, every two weeks for another 4 weeks, and one session in 3rd month.
  Interventions: Drug: Triamcinolone Hexacetonide; Device: Sham LED
- Experimental Group (Experimental): Transcutaneous PBM will be performed on the keloid in the preoperative period and on the remaining scar in the postoperative period using blue LED (470 nm, 0,4W, 24J per point on 10 linear points, total 240J). Frequency: Preoperative: every two weeks for 30 days. Postoperative: Immediately after surgery, weekly for 4 weeks, every two weeks for another 4 weeks, and one session in 3rd month.
  Intralesional administration of corticoid (IAC): intralesional injection of 20 mg/ml triamcinolone hexacetonide: two injections in the preoperative period with a two-week interval between injections and a monthly injection for three months in the postoperative period. The injections will be intralesional and will not surpass the dermis. The drug will be diluted with the same quantity of 2% lidocaine. The scar will be divided into equal parts of 1 cm² and the drug will be distributed equally, respecting the total dose per session of 20 mg for the face and 40 mg for other topographies.
  Interventions: Device: Photobiomodulation with blue led; Drug: Triamcinolone Hexacetonide

INTERVENTIONS:
Device: Photobiomodulation with blue led — Preoperative: every two weeks for 30 days. Postoperative: Immediately after surgery, weekly for 4 weeks, every two weeks for another 4 weeks, and one session in 3rd month. blue LED (470 nm, 0,4W, 24J per point on 10 linear points, total 240J).
  Arms: Experimental Group
Drug: Triamcinolone Hexacetonide — intralesional injection of 20 mg/ml. two injections in the preoperative period with a two-week interval between injections and a monthly injection for three months in the postoperative period. The injections will be intralesional and will not surpass the dermis. The drug will be diluted with the same quantity of 2% lidocaine. The scar will be divided into equal parts of 1 cm² and the drug will be distributed equally, respecting the total dose per session of 20 mg for the face and 40 mg for other topographies.
Device: Sham LED — A blue LED without power and biologic effect.
  Arms: Sham Group

SUMMARY:
A randomized, controlled, double-blind, clinical trial will be conducted to study the evaluate the effect of blue light combined with corticoid treatment in the preoperative and postoperative period of keloid removal surgery.

DETAILED DESCRIPTION:
Keloid scars are characterized by the excessive proliferation of fibroblasts and an imbalance between the production and degradation of collagen, leading to its buildup in the dermis. Although the genesis of this condition is not yet fully clarified, keloids are known to have a genetic component and are related to an increase in the expression of transforming growth factor beta (TGF-β). There is no "gold standard" treatment and recurrence is frequent. Therefore, novel treatment options are needed. In vitro studies have demonstrated that photobiomodulation (PBM) reduces the multiplication velocity and quantity of fibroblasts as well as the expression of TGF-β. This is a low-cost, noninvasive therapy with no side effects that has proved to be a good tool to complement the most established treatment. Therefore, the purpose of this study is to evaluate the effect of blue light combined with corticoid treatment in the preoperative and postoperative period of keloid removal surgery. A randomized, controlled, double-blind, clinical trial will be conducted involving two groups: 1) Sham (N = 29): intralesional administration of corticoid (IAC) and sham PBM in the preoperative and postoperative periods of keloid removal surgery; and 2) active PBM combined with IAC (N = 29) in the preoperative and postoperative periods of keloid removal surgery. Transcutaneous PBM will be performed on the keloid in the preoperative period and on the remaining scar in the postoperative period using blue LED (470 nm, 0,4W, 24J per point on 10 linear points, total 240J). The patients will answer two questionnaires: one for the assessment of quality of life (Qualifibro-UNIFESP) and one for the assessment of satisfaction with the scar (PSAQ). The team of plastic surgeons will answer the Vancouver Scar Scale (VSS). All questionnaires will be administered one, three, six, and twelve months postoperatively. The keloids will be molded in silicone prior to the onset of treatment and prior to excision to assess pre-treatment and post-treatment size. The same will be performed for the remaining scar at one, three, six, and twelve months postoperatively. The removed keloid will be sent for histopathological analysis for the determination of the quantity of fibroblasts, the organization and distribution of collagen (picrosirius staining), and the expression of TGF-β. All data will be submitted to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years;
* Fitzpatrick skin phototype I-VI;
* Keloid with no type of previous treatment;
* Recurring keloid after surgical excision;
* Recurring keloid after use of other therapies and at least three months without treatment.

Exclusion Criteria:

* Keloid in treatment;
* Pregnant and lactating women;
* Keloid with primary synthesis of the skin and no possibility of excision.
* Contraindications for undergoing surgery (e.g.: coagulopathies, diabetes myellitus, drug allergies);
* Contraindications for the use of corticosteroids;
* All types of Collagenosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
scar assessment by specialists (change in the scar of is being evaluated) | Baseline (after the clinical evaluation prior to the intervention) as well as one, three, six, and twelve months postoperatively.
  Blinded, calibrated, certified plastic surgeons will answer the Vancouver Scar Scale (VSS), which was translated into Portuguese by Santos et al. This scale focuses on four parameters:
  scar height and thickness, pliability, vascularity, and pigmentation to generate a score ranging from 0 to 13 points. The VSS set a precedent for the systematic evaluation of scars, taking a semiquantitative approach to organize a collection of subjective assessments.
Quality of Life of the patients (change in quality of life is being evaluated) | Baseline (after the clinical evaluation prior to the intervention) as well as one, three, six, and twelve months postoperatively.
  The Quality of Life of Patients with Keloid and Hypertrophic Scarring questionnaire. The participants will answer the questionnaires. Answer choices are on a Likert Scale with the following choices: -5 (totally inaccurate), -3 (inaccurate), -1 (somewhat inaccurate), 1 (fairly accurate), 3 (accurate), 5 (completely accurate).
patient satisfaction with the scar (change in the quality of scar is being evaluated) | Baseline (after the clinical evaluation prior to the intervention) as well as one, three, six, and twelve months postoperatively.
  The participants will also answer Part II (classification of satisfaction) of the Patient Scar Assessment Questionnaire (PSAQ) Participant answer: Very satisfied, Satisfied Dissatisfied and Very Dissatisfied.

SECONDARY OUTCOMES:
keloid and remaining scar size | These procedures will be performed in baseline (preoperatively) as well as one, three, six, and twelve months postoperatively.
  Molds will be made of the scars in light condensation silicone (Zhermack, Badia Polesine, Italy). The material will be stored in acrylic dishes and sent for analysis (optical coherence tomography) for the determination of area and volume.
Fibroblasts analysis | one time up to 4 weeks after preoperative treatment
  Quantitative analysis of the fibroblasts of the keloid specimens will be performed. For such, the histological slides with the samples will be stained with hematoxylin-eosin (H.E.). This analysis is to verify the number of fibroblasts only trough visual analysis.
analysis of collagen | one time up to 4 weeks after preoperative treatment
  analysis of collagen fibers will also be performed using additional slices stained with Picrosirius Red. This analysis is to verify the number of fibers of collagen and your organization only trough visual analysis.
analysis of TGF-β | one time up to 4 weeks after preoperative treatment
  and RNA extraction

CONTACTS AND LOCATIONS:
Overall Officials: Raquel AM Ferrari, Phd, Principal Investigator — Nove de Julho University (Uninove)
Locations (1):
- Nove de Julho University (Uninove), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pires JA, Bragato EF, Momolli M, Guerra MB, Neves LM, de Oliveira Bruscagnin MA, Ratto Tempestini Horliana AC, Porta Santos Fernandes K, Kalil Bussadori S, Agnelli Mesquita Ferrari R. Effect of the combination of photobiomodulation therapy and the intralesional administration of corticoid in the preoperative and postoperative periods of keloid surgery: A randomized, controlled, double-blind trial protocol study. PLoS One. 2022 Feb 15;17(2):e0263453. doi: 10.1371/journal.pone.0263453. eCollection 2022. PMID 35167583